CLINICAL TRIAL: NCT04465513
Title: A Randomized, Open-label, Parallel Study to Investigate the Efficacy of CARDIO Softgels PLUS Best-standard-of-care in the Recovery of Patients With COVID-19 Who Are Hospitalized as Well as Patients Following the Guidance From Public Health
Brief Title: Investigation of the Efficacy of CARDIO Softgels PLUS Best-standard-of-care in the Recovery of Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20CCHH
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-06

CONDITIONS: COVID; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Standard of Care + CARDIO (Active Comparator): Combination of CARDIO and Best Standard of Care
  Interventions: Dietary Supplement: Best Standard of Care + CARDIO
- Best Standard of Care (Placebo Comparator): Placebo and Best Standard of Care
  Interventions: Dietary Supplement: Best Standard of Care

INTERVENTIONS:
Dietary Supplement: Best Standard of Care + CARDIO — Combination of dietary supplement with clinical care
  Arms: Best Standard of Care + CARDIO
Dietary Supplement: Best Standard of Care — Combination of placebo with clinical care
  Arms: Best Standard of Care

SUMMARY:
Corona virus disease 2019 (COVID-19) is caused by SARS-CoV-2, a plus-sense single-stranded RNA virus. After an incubation period, which typically lasts for 5-6 days, COVID-19 patients present with a mild illness that lasts for a few days. Common symptoms are reminiscent of the flu, and include fever, dry cough and dyspnea. A large percentage of patients resolve the infection whereas others progress onto adult respiratory distress syndrome (ARDS) which impedes gas exchange between the alveolar space and the bloodstream and creates the need for assisted respiration. The objective of this study is to investigate the safety and efficacy of CARDIO supplementation in the recovery of those with COVID-19 infection following the guidance from public health by reducing the need for mechanical respiratory support, alleviating respiratory symptoms and reducing mortality.

DETAILED DESCRIPTION:
SARS-CoV-2, a plus-sense single-stranded RNA virus, is the etiologic agent of COVID-19. After an incubation period, which typically lasts for 5-6 days. COVID-19 patients present with a mild illness that lasts for a few days. Common symptoms are reminiscent of the flu, and include fever, dry cough and dyspnea. A large percentage of patients resolve the infection whereas others progress onto adult respiratory distress syndrome (ARDS) which impedes gas exchange between the alveolar space and the bloodstream and creates the need for assisted respiration.

It is estimated that between 5-10% of asthma patients do not respond to steroid-based therapies and require higher doses of medication to achieve control of their disease, or have asthma exacerbations, persistent symptoms and airway obstruction despite greater medication use. These steroid-resistant asthmatics typically have greater morbidity and disproportionately require 50-80% of asthma-related health care costs. The compromised state of the lung in steroid-resistant asthma patients is similar to former smoker patients, for which eosinophil presence in the lung is believed to be a major pro-inflammatory effector cell in the pathogenesis of asthma. Further, in the United States, chronic lung disease (primarily asthma) was the second most prevalent underlying condition in those admitted to hospital for COVID-19 infection in adults ages 18-49.

CARDIO is a safe, natural, salmon oil based, eosinophil effector function (EEF) reducing, softgel formulation. Fish oil, inclusive of salmon oil, or marine-derived omega-3 supplements have been established as cardioprotective. CARDIO has been studied in human clinical studies for the treatment of cardiovascular disease, and as an antioxidant, with an excellent safety record. CARDIO has demonstrated therapeutic potential for the treatment of allergic and inflammatory conditions, particularly those involving eosinophil effector functions. Specifically, CARDIO at 100 ug/ml inhibited eosinophil response to chemoattractant CCL11 in a Shape Change assay; inhibited eosinophil response to chemoattractant CCL11 in an integrin (CD11b) surface upregulation assay; and significantly enhanced apoptosis, in eosinophils sourced from immuno-modulated individuals. Previous studies have shown that fish oil reduces recruitment and infiltration of eosinophils into airways. Among the bioactive components in fish oil, it has been demonstrated that the docosahexaenoic acid (DHA) has an inhibitory effect on proliferation and migration of eosinophils. In vitro and animal dosing studies have been completed for therapeutic dose determination for an accelerated Phase 2 trial application.

Rationale:

Although the exact mechanism of action is unknown, based on in vitro and in vivo studies, it is hypothesized that CARDIO may reduce morbidity and mortality from COVID-19 by protecting respiratory epithelium and alveolar pneumocytes from eosinophil-mediated damage. In light of the mechanism of action outlined above, it is possible that CARDIO could be used as a therapeutic for COVID-19 with the goal of preventing progression into severe disease and in particular in preventing the need of a mechanical ventilation.

Study population:

The population being investigated are hospitalized patients, all with mild to moderate respiratory distress due to COVID-19. Though the age has a reasonably wide range to facilitate recruitment, the exclusions in place provide the required guidance measures to ensure patient safety and address associated comorbidities. Individuals most prone to SARS-CoV-2 and hospitalization as a result of SARS-CoV-2 infection are those with co-morbidities such as older age, cancer, cardiovascular disease and hypertension, type I or II diabetes, chronic obstructive pulmonary disease, obesity and on immunosuppressive treatments. Therefore, participants with the above co-morbidities will comprise the population of interest. However, in this context, each participant will be assessed on a case-by-case basis by the Qualified Investigator to ensure all inclusions and none of the exclusions are met, and that the safety of their participation in the study is critically evaluated. The requirement of mild to moderate COVID-19 will be assessed using the most up- to-date National Institutes of Health (NIH) Treatment Guidelines for the Clinical Presentation of People with SARS-CoV-2 Infection. Using the NIH guidelines for clinical presentation of COVID-19 and identification of mild and moderate disease severity will ensure potential patients are evaluated based on the most up-to-date information in the ever changing COVID-19 research landscape. The safety of patients will be assessed at each assessment day, a Data and Safety Monitoring Board will be established, and an interim analysis is planned to guide safe continuation of the study.

The objectives of this randomized, open-label study is to investigate the safety and efficacy of CARDIO plus best standard-of-care in reducing the need for mechanical respiratory support, alleviating respiratory symptoms and reducing mortality in patients with COVID-19 infection in patients who are hospitalized. The SPIRIT statement for protocols items for trials are followed and the reporting will be done in accordance with the Consolidated Standards of Reporting Trials (CONSORT) Statement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with signs and symptoms corresponding to COVID-19 viral infection and:
2. Admitted to hospital and who have been initiated with BSC treatment with mild to moderate disease as defined by the National Institutes of Health (NIH) Treatment Guidelines
3. Confirmation of COVID-19 infection This will be assessed by secondary laboratory confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) or comparable methodology used by the hospital from any diagnostic sampling - source for analysis and recovery
4. Males and females between 18 and 75 years of age, inclusive
5. Female patient is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
6. Willingness to complete assessments, questionnaires and records associated with the study
7. Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the study
2. Inability to take medications orally
3. Individuals with a known fish allergy or hypersensitivity reaction
4. Individuals with uncontrolled hypotension (systolic blood pressure < 90 mmHg) or need for vasopressor/inotropic medication
5. Individuals with renal impairment This will be assessed by increase of creatinine by 50% from baseline, glomerular filtration rate reduction by >25% from baseline or urine output of <0.5 ml/kg for 6 hours)
6. Individuals with gastrointestinal symptoms that require hospitalization (e.g. severe nausea, vomiting, diarrhea or/and abdominal pain) Any other condition, that, in the opinion of the QI, may adversely affect the patient's ability to complete the study or its measures or pose significant risk to the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring mechanical ventilator until end of study (Day 28) | Day 28
  Proportion of patients requiring mechanical ventilator until end-of-study, when comparing Best Standard of Care treatment (BSC) plus CARDIO unrefined salmon oil vs. BSC alone

SECONDARY OUTCOMES:
Clinical improvement | Day 10, Day 14, Day 28, or Day of discharge
  Clinical improvement assessed by the National Early Warning Score (NEWS) at Day 10, Day 14, Day 28 or day of discharge. Assessed by the National Early Warning Score (NEWS) which is a standardized tool that assesses disease severity and monitoring of patients in hospital. An aggregate score of respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness and temperature and the score is increased if supplemental oxygen is required. Each parameter is based on a scale of 0 - 3. 0=good, 3=poor
Clinical status | Day 10, Day 14, Day 28, or Day of discharge
  Clinical status assessed by the WHO Ordinal Scale for Clinical Improvement at Day 10, Day 14, Day 28 or day of discharge. Assessed by the WHO Ordinal Scale for Clinical Improvement which examines changes in clinical status and/or survival specific to COVID-19. This 8-point scale measures illness severity over time. 0 = no infection and 8 = dead
Time to clinical recovery | Day 28 or Day of discharge
  Time to clinical recovery, defined as normalization of fever, respiratory rate, oxygen saturation, and alleviation of cough, sustained for at least 72 hours, at Day 28 or day of discharge
Time to improvement in oxygenation for at least 48 hours | Day 28 or Day of discharge
  Time to improvement in oxygenation for at least 48 hours, defined by an increase in SpO2/FiO2 of 50 mmHg or greater compared to the nadir SpO2/FiO2, at Day 28 or day of discharge
Quality of life (QoL) | Day 0, Day 10, Day 14, and Day 28
  Quality of life assessed by the COVID-19 QoL questionnaire at Day 0, Day 10, Day 14, and Day 28. Assessed by the COVID-19 QoL questionnaire which asks questions about incident of different parameters related to deteriorating. It is on a scale of 1-5. 1=completely disagree, 5 = completely agree.
All-cause mortality | Day 28
  Death due to COVID-19 and other reasons
Duration of mechanical ventilator use until end-of-study (Day 28) | Day 28
  The difference between BSC plus CARDIO vs. BSC alone on duration of mechanical ventilator use until end-of-study
Oxygenation requirements assessed by oxygen saturation rates based on number of oxygenation free days during hospital stay | During hospital stay, on day of discharge if prior to Day 28, and on Day 28
  Oxygenation requirements during hospital stay, on day of discharge if prior to Day 28 and on Day 28, assessed by oxygen saturation rates based on number of oxygenation free days during hospital stay
Oxygenation requirements assessed by oxygen saturation rates based on incidence of new oxygen use, non-invasive ventilation or high flow oxygen devices | During hospital stay, on day of discharge if prior to Day 28, and on Day 28
  Oxygenation requirements during hospital stay, on day of discharge if prior to Day 28 and on Day 28, assessed by oxygen saturation rates based on incidence of new oxygen use, non-invasive ventilation or high flow oxygen devices
Oxygenation requirements assessed by oxygen saturation rates based on duration of new oxygen use, non-invasive ventilation or high flow oxygen devices | During hospital stay, on day of discharge if prior to Day 28, and on Day 28
  Oxygenation requirements during hospital stay, on day of discharge if prior to Day 28 and on Day 28, assessed by oxygen saturation rates based on duration of new oxygen use, non-invasive ventilation or high flow oxygen devices
Serial chest CT or X-ray findings | Day 10 and Day 28 or Day of discharge
  Serial chest CT or X-ray findings at Day 10, Day 28 or day of discharge
The number of days from hospital admission to hospital discharge | Up to Day 28
  The difference between BSC plus CARDIO vs. BSC alone on the number of days from hospital admission to hospital discharge
The total number of days on ventilator at Day 28 or day of discharge | Day 28 or Day of discharge
  The difference between BSC plus CARDIO vs. BSC alone on the total number of days on ventilator at Day 28 or day of discharge
The number of days in intensive care unit (ICU) at Day 28 or day of discharge | Day 28 or Day of discharge
  The difference between BSC plus CARDIO vs. BSC alone on the number of days in intensive care unit (ICU) at Day 28 or day of discharge
Temperature measurements after discharge and to end of study (Day 28) | Day 28 and after discharge
  The difference between BSC plus CARDIO vs. BSC alone on body temperature measurements after discharge and to end of study (Day 28)
Oxygen saturation measurements after discharge and to end of study (Day 28) | Day 28 and after discharge
  The difference between BSC plus CARDIO vs. BSC alone on oxygen saturation measurements after discharge and to end of study (Day 28). Oxygen saturation saturation measurements recorded using a pulse oximeter.
COVID-19 QoL measurements after discharge and to end of study (Day 28) | Day 28 and after discharge
  The difference between BSC plus CARDIO vs. BSC alone on COVID-19 QoL measurements after discharge and to end of study (Day 28). Quality of life assessed by the COVID-19 QoL questionnaire which asks questions about incident of different parameters related to deteriorating. It is on a scale of 1-5. 1=completely disagree, 5 = completely agree.

OTHER OUTCOMES:
Adverse Events | Day 0 and up to day 28
  Incidence of pre-emergent and post-emergent adverse events (AEs) and serious adverse events (SAEs) during the 28 days of supplementation or until day of discharge and during home follow up
Blood pressure | Day 0 and up to day 28
  Systolic and diastolic blood pressure values for the CARDIO softgel + BSC group will be compared with those of the BSC group during the 28-day supplementation period or until day of discharge and during home follow up
Heart rate | Day 0 and up to day 28
  Heart rate values for the CARDIO softgel + BSC group will be compared with those of the BSC group during the 28-day supplementation period or until day of discharge and during home follow up
Abnormality in laboratory tests | Day 28 or Day of discharge
  Frequency of clinically significant laboratory abnormalities at Day 28 or day of discharge
Body mass Index (BMI) | Day 0, Day 10, Day 14, and Day 28 from baseline
  BMI values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Complete blood count (CBC) | Day 0, Day 10, Day 14, and Day 28 from baseline
  CBC values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Aspartate transaminase (AST) | Day 0, Day 10, Day 14, and Day 28 from baseline
  AST values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Alanine transaminase (ALT) | Day 0, Day 10, Day 14, and Day 28 from baseline
  ALT values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Alkaline phosphatase (ALP) | Day 0, Day 10, Day 14, and Day 28 from baseline
  ALP values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Bilirubin | Day 0, Day 10, Day 14, and Day 28 from baseline
  Bilirubin values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Sodium ion | Day 0, Day 10, Day 14, and Day 28 from baseline
  Sodium ion values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Potassium ion | Day 0, Day 10, Day 14, and Day 28 from baseline
  Potassium ion values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Chloride ion | Day 0, Day 10, Day 14, and Day 28 from baseline
  Chloride ion values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Creatinine | Day 0, Day 10, Day 14, and Day 28 from baseline
  Creatinine values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
eGFR | Day 0, Day 10, Day 14, and Day 28 from baseline
  eGFR values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
HbA1c | Day 0, Day 10, Day 14, and Day 28 from baseline
  HbA1c values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
Glucose | Day 0, Day 10, Day 14, and Day 28 from baseline
  eGFR values for the CARDIO softgel + BSC group will be compared with those of the BSC group using statistical analysis to determine significant difference between the two groups. Samples are taken in the days stated below.
C-Reactive protein (CRP) | Day 0, Day 10, Day 14, and Day 28 from baseline
  Changes in CRP from screening

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (8):
- Brazil (3):
  - Hospital Universitario Cassiano Antonio de Morais, Vitória, Espírito Santo
  - - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Instituto Santa Marta de Ensino e Pesquisa, Taguatinga
- KGK Science Inc., London, Ontario, Canada
- Hungary (2):
  - Markhot Ferenc Oktatókórház és Rendelőintézet, Eger, Eger
  - Albert Schweitzer Kórház-Rendelőintézet, Hatvan, Hatvan
- The American British Cowdray Medical Center I.A.P., Mexico City, Mexico
- General Hospital Paracin, Paraćin, Serbia

IPD SHARING:
Plan to Share IPD: No